CLINICAL TRIAL: NCT04980781
Title: Evaluation of the Implementation of a New Therapy for Bulimia Nervosa and Binge Eating Disorder; Physical Exercise and Dietary Therapy (PED-t), in a Naturalistic Setting
Brief Title: Evaluation of the Implementation of PED-t in a Naturalistic Setting
Acronym: EVA-PEDt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Collaborators: Norwegian School of Sport Sciences (Other); University of Tromso (Other); The Norwegian Women´s Public Health Association (Other); Norwegian Council for Mental Health (Other); The Dam Foundation (Other); The Vibeke Skofterud Foundation (Unknown)
Responsible Party: Principal Investigator, Therese Fostervold Mathisen, Associate professor, Ostfold University College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 40503
Record Dates: First submitted 2021-03-22; First posted 2021-07-28 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder
Keywords: remission; treatment; therapy; physical exercise; dietary therapy; diet; physical activity; naturalistic; Exercise referral centers; Healthy Living Centers; eating disorders; implementation
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Motor Activity; Feeding and Eating Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Employees and management in a ECR receive training in PED-t, and successively arrange the therapy. Experiences with the program training, and expectations to and experiences from giving the therapy, are the main research questions. Managements will be interviewed according to experiences with management of- and suitability of the therapy in the ECR
  Eligible participants with bulimia nervosa or binge eating disorder are recruited for therapy in the ECR. Their expectations to- and experiences from having therapy in the ECR are the main research questions, in addition to evaluation of therapy success.
  A previous RCT has evaluated the treatment efficiency by comparing it to a control group and another standardized treatment intervention. As such, the main focus of the current study is to evaluate experiences from arranging PED-t in a naturalistic setting, and secondly to evaluate if treatment efficiency can be replicated.
Masking Description: No masking, as this is a non-controlled intervention trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving PED-t (Experimental): Participants, i.e. females with bulimia nervosa or binge eating disorder, are recruited for therapy in the trained ERC. The treatment program consists of 20 behavioral therapy sessions covering 16 weeks, and with single follow-up sessions at 2-, and 4- months post-therapy.
  Participants are interviewed on the expectations to- and experiences from having therapy in the ECR, and monitored and evaluated on therapy effectiveness (i.e. diagnostic outcomes).
  Interventions: Behavioral: Physical exercise and dietary therapy (PED-t)
- Therapists and management in ERC offering PED-t (Experimental): Employees in the ECR and the management will be trained in giving PED-t in their facility, and will then perform therapy with a single group of participants recruited.
  Therapists/employees trained in PED-t will be interviewed about their expectations to- and experiences from giving the PED-t, and also being monitored according to therapy manual fidelity.
  The management at the facility offering PED-t will be interviewed about their experiences on administration and implementation of the PED-t in their facility.
  Interventions: Procedure: Implementation program for PED-t in ERC

INTERVENTIONS:
Behavioral: Physical exercise and dietary therapy (PED-t) — Behavioral therapy: Physical exercise and dietary therapy (PED-t) is a treatment of bulimia nervosa and binge eating disorder, relying on guided, progressive resistance exercise therapy and dietary therapy (dietary education and group discussions) following a designed therapy manual.
  Other Names: PED-t; FAKT
  Arms: Participants receiving PED-t
Procedure: Implementation program for PED-t in ERC — Participating in a training program for therapists in PED-t; to increase knowledge of eating disorders and to be able to implement and run the PED-t. Training program consists of a therapy manual, digital lectures, and 3 work shops.
  Arms: Therapists and management in ERC offering PED-t

SUMMARY:
The Eva-PED-t project will evaluate implementation of a new therapy for eating disorders, called PED-t (Physical Exercise and Dietary therapy), in a new treatment arena for such illnesses. By this, Eva-PED-t evaluates effectiveness- and efficacy outcomes, with the latter highlighting both the user-, the therapists- and the management perspectives. The research group behind this initiative comprises the founders of the PED-t, and holds extensive expertise on research methodology, eating disorders, health science, and exercise medicine, affiliated high-ranked research-intensive universities. Previous documentation of poor implementation of evidence-based knowledge in public health services reveal poor or no translation of new research findings for improved screening, treatment or medical procedures into real life settings. This may impair public health service outcomes, as less effective or ineffective treatment or procedures are routinely preferred. In a randomized controlled trial, the Eva-PED-t partnership recently found a new therapy for eating disorders (PED-t) to be comparable effective to the currently recommended treatment (NCT02079935). Specific advantages with PED-t, are the use of professionals not currently used in therapy of mental disorders, and the efficiency of arranging therapy in groups, hence effectively dealing with the high request for therapy. The Eva PED-t collaborative is motivated by the knowledge of high prevalence of mental illnesses, for which there is a need to improve treatment access and -efficiency. Adding to this scenario, is the new and more prevalent diagnosis of eating disorders, binge eating disorder, for which specialized health services have no prioritization for treatment. Addressing requirements for improved therapy access demands investigation of new treatments and new ways of delivery. The PED-t responds to this request, still recommendation for a broad implementation necessitate exploration of implementation strategies and experiences.

DETAILED DESCRIPTION:
Implementation research intends to identify facilitating and obstructing elements in the process of transferring evidence-based practices from controlled settings to naturalistic settings. Unfortunately, the implementation of evidence-based knowledge is challenged by lack of institutional resources and insufficient prioritization by the management, and lack of prioritization by funders and academic researchers. As such, a lag time before evidence-based knowledge from research is translated in to real world practice is typically estimated to be about 14-20 years. The delay in implementation of evidence-based practice is found to be specifically relevant in health care services, hence, ultimately depriving patients from best practice. Exercise referral centers (ERC, also known as Healthy Living Centers) are part of the municipally public health care, providing support for improved healthy living behavior. Service users are confident by the professional skills in the ERC, and trust the service to be evidence-based. However, there are a wide variety in program approaches and methodology, most with no evidence-based foundation, and a lack of documentation on effects. Hence originally, the UK National Institute for Health and Clinical Excellence (NICE) recommended not to commission ERC in primary health care other than in well-designed research studies. The ERC's are in an early progress, still exploring their role in public health care and having stakeholders requesting evidence-based methods, and as such, identification of successful interventions at the ERC's is necessitated.

The Eva-PED-t has the potential to pick up on the shortfalls in documentation of effectiveness outcomes and exploration of efficacy of evidence-based interventions at the ERC's, and the poor implementation of evidence-based treatment in public health services in general. The EVA_PED intend to evaluate the implementation of the PED-t in the public health care services ERC in terms of effectiveness and efficacy, and by a mixed methods design. By relying on the original team behind the development of the PED-t to train the therapists, inform and supervise the management, and to provide support during implementation, this project has the potential to ease the implementation process. As such, the EVA-PED aim to follow the request to evaluate the total implementation success (i.e. the sum of the effectiveness of treatment and the experiences of implementation within the organization).

The researchers behind the EVA-PED finalized the evaluation of effectivity from PED-t on treatment of eating disorders in 2018 (NCT02079935), bringing optimism on increased therapy access, lowering barriers for treatment seeking behavior, and facilitating a more effective treatment delivery. Having the PED-t research team initiating Eva-PED-t, this project will bypass the delay in translation of evidence-based knowledge to real life settings. The Eva-PED-t has the potential to identify any elements undermining optimal uptake of this evidence-based treatment in public health services. Informed on previous challenges on successful implementation of evidence-based procedures, Eva-PED-t grasp on these most critical elements. Providing practical training and adequate time for preparations, mentoring during therapy operation, relying on therapy elements similar to what the therapists have practiced in their regular work, and by communicating, involving and motivating several levels in the organizations (management and therapists); the EVA_PED target the most critical elements previously found to impair successful implementation. Additionally, by involving former patients and therapists from the PED-t intervention as user groups, combined with the findings from in depth interviews in the corresponding groups of patients and therapists, the EVA-PED will evaluate adjustments of the therapy and arrangement according to their experiences and advices.

The EVA-PED-t project aims to evaluate the success of adopting and operating the evidence-based PED-t in naturalistic settings like ERC's, physiotherapy clinics and multidisciplinary medical centers. By this, the project intends to study effectiveness outcomes and efficacy outcomes, with the latter highlighting both the user perspectives, the therapists- and the management perspectives. A part of the efficacy outcomes, is evaluation on the treatment fidelity by individual therapists.

This generate the following main- and secondary research questions (RQ):

Main RQ:

1. Which elements promotes or discourages the implementation of PED-t according to; a) the therapists, and b) the management at the therapy cites?

Secondary RQ's:

1. How well is the implementation quality concerning treatment fidelity in a naturalistic setting?
2. What are the experiences amongst the patients receiving PED-t in a naturalistic setting?
3. How effective is the PED-t in a naturalistic setting, evaluated in remission from diagnosis, in rating of quality of life, in intensity of symptoms for depression, anxiety and symptoms of an eating disorder, and in changes of eating- and exercise behavior?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bulimia nervosa or binge eating disorder
* BMI 17.5 - 40
* Women

Exclusion Criteria:

* Being/planning to become pregnant during the therapy period
* Competitive athlete
* Concurrent severe symptom- or personality disorder in need of other treatment options

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Expectations and readiness for running the PED-t (therapists) | 1 hour in June 2021, pre-therapy
  After training for PED-t; what are the therapists expectations to offering the PED-t and how able and ready do they feel about taking care of the patients? (semistructured interviews)
Experiences after running the PED-t (therapists) | 1 hour in December 2021, post-therapy
  After running the PED-t; what are the therapists experiences from offering the PED-t and (semistructured interviews)
Expectations on receiving PED-t in the ERC (patients) | 1 hour in August 2021, pre-therapy
  What are the patients expectations to receive PED-t in in the ERC? (semistructured interviews)
Experiences from receiving PED-t in the ERC (patients) | 1 hour in December 2021, post-therapy
  What are the patients experiences from receiving PED-t in in the ERC? (semistructured interviews)
Management of training program and therapy in the ERC (leaders in the ERC) | 1 hour in August 2021, pre-therapy
  What are the leaders experiences on managing therapy training for employees, and expectations to offer a new therapy in the local ERC? (semistructured interviews)
Management/implementation of PED-t in the ERC (leaders in the ERC) | 1 hour in December 2021, post-therapy
  What are the leaders experiences on managing/implementing the PED-t in the local ERC? (semistructured interviews)

SECONDARY OUTCOMES:
Therapy manual fidelity | Once per 16 weeks (August-December)
  Electronic questionnaire measuring therapy manual fidelity, distributed on a weekly basis. Responding yes/no to whether specific topics has been addressed.
Rating of life quality before therapy | Pre-therapy, week 0
  QoL measured with the Satisfaction with life scale. This is a short 5-item scale measuring overall contentment with life compared to personal standards and expectations, using a 5-point Likert scale ranging from1 (never true) to 7 (always true) (Diener, 1994)
Rating of life quality after therapy | Post-therapy, week 17
  QoL measured with the Satisfaction with life scale. This is a short 5-item scale measuring overall contentment with life compared to personal standards and expectations, using a 5-point Likert scale ranging from1 (never true) to 7 (always true) (Diener, 1994)
Symptoms of depression before therapy | Pre-therapy, week 0
  Measured with the Beck Depression Inventory. Consists of 22 items rated from 0 to 3, resulting in a total score up to 65 points, and where scoring of 21 or above indicates having symptoms of depression.
Symptoms of depression after therapy | Post-therapy, week 17
  Measured with the Beck Depression Inventory. Consists of 22 items rated from 0 to 3 (one item scores 0-1), resulting in a total score up to 64 points, in which higher scoring means higher severity, and where scoring of 21 or above indicates having symptoms of depression.
Symptoms of anxiety before therapy | Pre-therapy, week 0
  Measured with the Beck Anxiety Inventory. Consists of 21 items, scored from 0-3, with higher scoring indicating higher severity.
Symptoms of anxiety after therapy | Post-therapy, week 17
  Measured with the Beck Anxiety Inventory. Consists of 21 items, scored from 0-3, with higher scoring indicating higher severity.
Symptoms of compulsive exercise before therapy | Pre-therapy, week 0
  Measured with the Compulsive exercise test. CET is a 24-item instrument scored on a 5-point Likert scale (0 = never true, 5 = always true), and evaluated with five different subscale mean scores.
Symptoms of compulsive exercise after therapy | Post-therapy, week 17
  Measured with the Compulsive exercise test. CET is a 24-item instrument scored on a 5-point Likert scale (0 = never true, 5 = always true), and evaluated with five different subscale mean scores.
Symptoms of eating disorder before therapy | Pre-therapy, week 0
  Evaluated by the Eating Disorder Examination questionnaire. Consists of 28 items, for which 22 items are rated from 0-6, and 6 items consists of selfreported number of binge-eating or purging episodes. Higher items scorings means higher severity, a total score above 2.5 indicates a diagnosis of eating disorder (according to validation in a Norwegian sample), and diagnosis necessitates at least 1 episode of binge-eating and/or purging per week.
Symptoms of eating disorder after therapy | Post-therapy, week 17
  Evaluated by the Eating Disorder Examination questionnaire. Consists of 28 items, for which 22 items are rated from 0-6, and 6 items consists of selfreported number of binge-eating or purging episodes. Higher items scorings means higher severity, a total score above 2.5 indicates a diagnosis of eating disorder (according to validation in a Norwegian sample), and diagnosis necessitates at least 1 episode of binge-eating and/or purging per week.
Evaluation of an eating disorder diagnosis | Pre-therapy, week 0
  Evaluation on diagnosis by the Eating Disorder Examination questionnaire (EDE-q) and clinical interview to manually affirm symptoms reported in EDE-q.
How effective is the PED-t in a naturalistic setting, evaluated in remission from diagnosis? | Post-therapy, week 17
  Evaluation on diagnosis by the Eating Disorder Examination questionnaire (EDE-q) and clinical interview to manually affirm symptoms reported in EDE-q.
Symptoms of eating disorder behavior | Once per week during 16 weeks of therapy
  Selfreported number of binge-eating episodes and purging episodes per week.

OTHER OUTCOMES:
Cardiorespiratory fitness (CRF) in patients before therapy | Pre-therapy, week 0
  CRF will be measured by performing a cardiopulmonary exercise test on a treadmill (ELG 90/200 Sports; Woodway, Weil am Rhein, Germany) with an incremental modified Balke protocol until exhaustion (Edvardsen,Hem, & Anderssen, 2014). Results are presented as ml oxygen consumed per kg bodymass per minute. Valid test requires measures of respiratory exchange ratio (RER) above 1.10, and lactate concentration above 7.0 mmol/L measured 1 min after test termination. A Borg scale rating above 17 may support evaluation if needed.
Cardiorespiratory fitness (CRF) in patients after therapy | Post-therapy, week 17
  CRF will be measured by performing a cardiopulmonary exercise test on a treadmill (ELG 90/200 Sports; Woodway, Weil am Rhein, Germany) with an incremental modified Balke protocol until exhaustion (Edvardsen,Hem, & Anderssen, 2014). Results are presented as ml oxygen consumed per kg bodymass per minute. Valid test requires measures of respiratory exchange ratio (RER) above 1.10, and lactate concentration above 7.0 mmol/L measured 1 min after test termination. A Borg scale rating above 17 may support evaluation if needed.
Resting metabolic rate (RMR) in patients before therapy | Pre-therapy, week 0
  RMR will be measured by performing indirect calorimetry; 20 minutes in total. A valid RMR (kcal per day) will be defined according to the current recommendation emphasizing the importance of a SS, being defined as 5 min periods with less than 10% CV for VO2 and VCO2.
Resting metabolic rate (RMR) in patients after therapy | Post-therapy, week 17
  RMR will be measured by performing indirect calorimetry; 20 minutes in total. A valid RMR (kcal per day) will be defined according to the current recommendation emphasizing the importance of a SS, being defined as 5 min periods with less than 10% CV for VO2 and VCO2.
Blood pressure in patients before therapy | Pre-therapy, week 0
  Resting blood pressure (systolic and diastolic) will be measured twice according to a standardized protocol (Mancia et al., 2013) with an automatic blood pressure device (Spot Vital Signs LXi; Welch Allyn, Skaneateles Falls, NY).
Blood pressure in patients after therapy | Post-therapy, week 17
  Resting blood pressure (systolic and diastolic) will be measured twice according to a standardized protocol (Mancia et al., 2013) with an automatic blood pressure device (Spot Vital Signs LXi; Welch Allyn,Skaneateles Falls, NY).
Body composition (muscle mass) in patients before therapy | Pre-therapy, week 0
  Body composition (i.e. muscle mass in kilogram, kg) will be measured by DXA.
Body composition (bone mass) in patients before therapy | Pre-therapy, week 0
  Body composition (i.e. bone mineral density in gram) will be measured by DXA.
Body composition (visceral adipose tissue) in patients before therapy | Pre-therapy, week 0
  Body composition (i.e. visceral adipose tissue in gram) will be measured by DXA.
Body composition (fat mass) in patients before therapy | Pre-therapy, week 0
  Body composition (i.e. fat mass in kilogram, kg, and percent, %, of total body mass) will be measured by DXA
Body composition (muscle mass) in patients after therapy | Post-therapy, week 17
  Body composition (i.e. muscle mass in kilogram, kg) will be measured by DXA.
Body composition (bone mass) in patients after therapy | Post-therapy, week 17
  Body composition (i.e. bone mineral density in gram) will be measured by DXA.
Body composition (visceral adipose tissue) in patients after therapy | Post-therapy, week 17
  Body composition (i.e. visceral adipose tissue in gram) will be measured by DXA.
Body composition (fat mass) in patients after therapy | Post-therapy, week 17
  Body composition (i.e. fat mass in kilogram, kg, and percent, %, of total body mass) will be measured by DXA.
Level of Physical activity in patients before therapy | Pre-therapy, week 0
  Level of physical activity will be measured by Aktigraph for 7 consecutive days using the ActiGraph accelerometer (ActiGraph GT3x; Actigraph, LCC, Pensacola, FL) placed on their right hip. Results are given as counts per minute, and will be compared to national representative results.
Level of Physical activity in patients after therapy | Post-therapy, week 17
  Level of physical activity will be measured by Aktigraph for 7 consecutive days using the ActiGraph accelerometer (ActiGraph GT3x; Actigraph, LCC, Pensacola, FL) placed on their right hip. Results are given as counts per minute, and will be compared to national representative results.
OSTRC Questionnaire for physical health issues | Once weekly during 16 weeks of therapy
  Questionnaire developed to capture any illness or injuries depriving patients from weekly exercise sessions. Any episode is reported, and number of days with no exercise is given together with anatomical localization.

CONTACTS AND LOCATIONS:
Overall Officials: Therese F Mathisen, PhD, Principal Investigator — Faculty of Health and Welfare, Østfold University College
Locations (1):
- Fredrikstad Frisklivssentral (Exercise Referal Center in the municipality of Fredrikstad), Fredrikstad, Norway

IPD SHARING:
Plan to Share IPD: No
Data is reserved the research group

REFERENCES:
- [Background] Mathisen TF, Rosenvinge JH, Pettersen G, Friborg O, Vrabel K, Bratland-Sanda S, Svendsen M, Stensrud T, Bakland M, Wynn R, Sundgot-Borgen J. The PED-t trial protocol: The effect of physical exercise -and dietary therapy compared with cognitive behavior therapy in treatment of bulimia nervosa and binge eating disorder. BMC Psychiatry. 2017 May 12;17(1):180. doi: 10.1186/s12888-017-1312-4. PMID 28494809